CLINICAL TRIAL: NCT06613438
Title: The Effect of Non-Invasive Electrical Stimulation Therapy on Gastroesophageal Reflux Disease (GERD)
Brief Title: Safety and Effectiveness of eGERD Device to Reduce Gastroesophageal Reflux Disease (GERD) Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gerd Care Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-PRO-0300; MOH_2024-05-12_013278 (Registry Identifier: MyTrial (Israel Ministry of Health Clinical Trial Registry))
Record Dates: First submitted 2024-09-18; First posted 2024-09-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-09

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
Keywords: Electrostimulation; Refulx; Regurgitation; eGERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active (Experimental): Participants in the active arm will be using a functional version of the investigational device for 28 days.
  Interventions: Device: eGERD device
- Control (Sham Comparator): Participants in the control arm will be using a sham version of the investigational device for 28 days.
  Interventions: Device: eGERD_Sham

INTERVENTIONS:
Device: eGERD device — The eGERD device is a novel device developed by GerdCare Medical for reducing symptoms of GERD. The device is noninvasive and designed for self-use in the home environment. It is applied on the abdominal skin and generates electrical stimulation pulses.
  For optimized effect, the stimulation is synchronized with the breathing phase, such that it is active mainly during inhalation. The stimulation intensity can be adjusted by the user.
  Arms: Active
Device: eGERD_Sham — The eGERD_Sham is a sham version of the eGERD device. It is capable of inducing sensation of electrical stimulation pulses in the target abdominal muscles without a therapeutic effect. Aside from this difference, the eGERD_Sham is identical to the eGERD device.
  Arms: Control

SUMMARY:
The purpose of this research is to evaluate the safety and effectiveness of the eGERD device, which is a novel device for treating Gastroesophageal Reflux Disease (GERD).

The main questions this research aims to answer are:

1. Does the eGERD device reduce acidity in the esophagus?
2. Does the eGERD device reduce GERD symptoms such as heartburn and regurgitation?
3. What medical problems do participants have when using the eGERD device?

To assess the acidity in the esophagus, a wireless standard-of-care capsule called Bravo will be placed in the participants esophagus (throat) for several days.

To assess GERD symptoms, participants will be requested to report symptoms they experience using a smartphone application.

Researchers will compare a real version of the eGERD device to a sham version (a look-alike device that has no therapeutic effect) to see if the eGERD device is effective in treating GERD.

DETAILED DESCRIPTION:
The study includes two consecutive phases: a 14-day washout phase followed by a 28-day device treatment phase.

The washout phase starts on or shortly after the Screening visit, in which the participants sign the informed consent form (ICF) and their eligibility criteria are assessed. The first day of the washout phase is considered Day 1 of the study.

In the washout phase, participants are instructed to avoid any GERD-treatment medications (including antacids), either prescribed or over-the-counter (OTC), and to keep their regular daily routines.

Participants are also instructed to report occurrence and severity of GERD-related symptoms using the eGERD smartphone application.

GERD-HRQL questionnaire are filled at the onset (Day 1) and at the end (Day 14) of this phase. Questionnaire score obtained at the end of the washout phase (QoL Score baseline) are regarded as baseline for the QoL secondary endpoint.

On the last day of the washout phase (Day 14), a 24h wireless pH monitoring test (Bravo) is initiated, in order to obtain acid exposure time (AET) and DeMeester score (DM) baseline levels.

The device treatment phase consists of continuous usage of the study device for 28 days.

At the onset of the device treatment phase, the pH monitoring data is downloaded and analyzed, to establish AET and DM baseline levels. To be eligible for randomization and study device usage, a participant must have (i) at least 18 hours of baseline monitoring data , and (ii) abnormal baseline AET (above 6%). Ineligible subjects are classified as screen failures. participants with insufficient baseline monitoring data (less than 18 monitoring hours) are offered to extend the baseline monitoring for another 24 hours.

Upon establishing participant eligibility and performing randomization, a new 96h wireless pH monitoring test is initiated using the same Bravo capsule already in place. At the same time, the participant starts using the study device. One day later, a short clinic visit is held in which proper operation of the study device is verified. At the end of the 96h pH monitoring test, the monitoring system is collected and the data downloaded.

Usage of the study device is continued from randomization for 28 days. Esophageal acid exposure time (AET) and DeMeester score (DM) obtained from the 24h wireless pH monitoring test are regarded as baseline for AET primary endpoint and DeMeester score secondary endpoint, respectively.

Esophageal acid exposure time and DeMeester score obtained from the last Complete Monitoring Day of the 96h monitoring test are considered AET primary endpoint and DeMeester score secondary endpoint, respectively.

Throughout this phase, participants are using a study device (either functional or sham), after receiving instructions on its usage. Participants are instructed to use the study device 24 hours per day, 7 days per week (excluding device charging, bathing, sporting, private situations, etc.).

Usage of antacids (Gaviscon Regular Strength antacid tablets, 2-4 tablets, up to 4 times a day) as a rescue treatment is allowed after the Bravo system has been collected from the participant (Day 19). Rescue treatment usage is reported and recorded. Usage of any other type of GERD-treatment is prohibited throughout the entire phase.

GERD-HRQL questionnaire is filled at the end of this phase (or on end-of-study visit, in case of early termination). Resulting score is regarded as QoL secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 22 - 75
* Has been typically suffering from at least three heartburn and/or regurgitation episodes per week during the past three months.
* Undergone a wireless (Bravo) pH monitoring test during the past 24 months prior to enrollment into the current study, following a 7-day (min.) off-PPI period, with AET ≥6% (as defined in section 7.2) in at least 2 monitoring days AND when averaged over all monitoring days of the test; or Undergone a catheter-based pH monitoring test during the past 24 months prior to enrollment into the current study, following a 7-day (min.) off-PPI period, with AET ≥6% (as defined in section 7.2).
* Able and willing to give informed consent for participation in the study and to comply with all study requirements, including operating the smartphone application.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Previously undergoing gastric or esophageal surgery
* Active peptic ulcer disease
* Esophageal or gastric varices or esophageal peptic stricture
* Severe dysphagia
* History of suspected or confirmed esophageal or gastric cancer
* History of any other malignancy in the last 2 years
* Pregnant women or women intending to become pregnant during the trial period
* Uncontrolled diabetes mellitus, defined as HbA1c > 7.5%
* Severe cardiac conditions such as cardiac arrhythmia or ischemia or cardiac pacemaker / defibrillator
* Having any implanted electrical device (e.g. sacral nerve stimulation, brain stimulator, others)
* Known allergy to the device's adhesives/patches
* Severe pulmonary diseases
* History of significant multisystem diseases (e.g. kidney failure, liver failure)
* Known autoimmune or a connective tissue disorder (e.g. scleroderma, CREST-syndrome, Sjogren's Syndrome), requiring therapy in the preceding 2 years
* History of Barrett's esophagus
* Para-esophageal hiatal hernia
* Known history of sliding hiatal hernia ≥4 cm in the last 3 years
* Known history of erosive esophagitis Grade C or D (LA classification) in the past 5 years
* Obesity, defined as BMI>32
* History of gastroparesis
* History of fibromyalgia, epilepsy, endometriosis
* Umbilical hernia >3cm
* Past usage experience with the study device
* Those currently enrolled in any other interventional clinical study
* Inability to sign the informed consent
* Inability to understand and fill the reports and questionnaires included in the study
* Inability to follow the study requisites
* Other medical conditions/medications that would interfere with subject safety or data collection in the opinion of the PI

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number and severity of Adverse Device Effects (ADEs) | From the beginning (Day 15) to the end (Day 42) of the device treatment phase
  Number and severity of Adverse Device Effects (ADEs) occurring when using the investigational device.
Change in esophageal acid exposure time | First pH monitoring day (Day 15) and last pH monitoring day (Day 19)
  Magnitude of change (from baseline to within normal limits) of acid exposure time (AET), as measured in a wireless pH monitoring test (Bravo™) conducted following a 14-day washout phase.

SECONDARY OUTCOMES:
Usage of rescue treatment | From the end of the pH monitoring test (Day 19) to the end of the device treatment phase (Day 42)
  The daily number of reported rescue treatment events, averaged over the period allowed for rescue treatment
Number of subjects electing to withdraw their consent | From the beginning (Day 15) to the end (Day 42) of the device treatment phase
  Number of subjects electing to withdraw their consent during the device treatment phase
Quality of life improvement | End of the washout phase (Day 14) and end of the device treatment phase (Day 42)
  Magnitude of change (from baseline) of the total score obtained in GERD-HRQL (GERD Health-Related Quality of Life) questionnaire.
Change in DeMeester Score | First pH monitoring day (Day 15) and last pH monitoring day (Day 19)
  Magnitude of change (from baseline to within normal limits) of DeMeester score, as measured in a wireless pH monitoring test (Bravo™) conducted following a 14-day washout phase.
Change in the frequency of regurgitation events | End of the washout phase (Day 14) and end of the device treatment phase (Day 42)
  Magnitude of change in the frequency of regurgitation events reported by patients using the smartphone application, when averaged over the last week of the device treatment phase, compared to the last week of the washout phase
Change in the frequency of heartburn events | End of the washout phase (Day 14) and end of the device treatment phase (Day 42)
  Magnitude of change in the frequency of heartburn events reported by patients using the smartphone application, when averaged over the last week of the device treatment phase, compared to the last week of the washout phase

OTHER OUTCOMES:
Change in esophageal acid exposure time (absolute) | First pH monitoring day (Day 15) and last pH monitoring day (Day 19)
  Magnitude of absolute change (from baseline) of acid exposure time (AET), as measured in a wireless pH monitoring test (Bravo™) conducted following a 14-day washout phase.
Change in DeMeester Score (absolute) | First pH monitoring day (Day 15) and last pH monitoring day (Day 19)
  Magnitude of absolute change (from baseline) of DeMeester score, as measured in a wireless pH monitoring test (Bravo™) conducted following a 14-day washout phase.

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Gastroenterology department, Emek medical center (EMC), Afula
  - Gastroenterology department, Rambam Health Care Campus, Haifa
  - Gastroenterology department, Rabin medical center (RMC), Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.gerd-care.com/join-our-clinical-study